CLINICAL TRIAL: NCT02563769
Title: Phase 1, Double-Blind, Placebo-Controlled Assessment of Potential Interactions Between Intravenous Cocaine and Clavulanic Acid
Brief Title: Clavulanic Acid (CLAV) and Cocaine Interaction Safety Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 23222; 1U54DA039002-01 (NIH)
Record Dates: First submitted 2015-08-06; First posted 2015-09-30 (Estimated); Results first posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Cocaine Dependence; Cocaine Addiction; Cocaine Abuse; Cocaine-Related Disorders
Keywords: Cocaine; Clavulanic Acid
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Clavulanic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Clavulanic Acid (CLAV) 250mg; CLAV 500mg then Placebo (PBO) (Experimental): Clavulanic acid OR Placebo to be given in combination with intravenous cocaine; Day #2: Clavulanic Acid 250 mg (low dose); Day #3: Clavulanic Acid 500 mg; Day #4: Placebo
  Interventions: Drug: Clavulanic acid; Drug: Intravenous cocaine; Drug: Placebo
- CLAV 250mg; PBO; then CLAV 500mg (Experimental): Clavulanic acid OR Placebo to be given in combination with intravenous cocaine; Day #2: Clavulanic Acid 250 mg (low dose); Day #3: Placebo; Day #4: Clavulanic Acid 500 mg
  Interventions: Drug: Clavulanic acid; Drug: Intravenous cocaine; Drug: Placebo
- PBO; CLAV 250mg; then CLAV 500mg (Experimental): Clavulanic acid OR Placebo to be given in combination with intravenous cocaine; Day #2: Placebo; Day #3: Clavulanic Acid 250 mg (low dose); Day #4: Clavulanic Acid 500 mg
  Interventions: Drug: Clavulanic acid; Drug: Intravenous cocaine; Drug: Placebo

INTERVENTIONS:
Drug: Clavulanic acid — Clavulanic acid will be administered orally in 250mg capsules
  Other Names: CLAV
Drug: Intravenous cocaine — 20/40mg Cocaine will be administered by IV
  Other Names: Coc
Drug: Placebo — Placebo will be administered orally in capsules identical to CLAV and be filled with crystalline microcellulose
  Other Names: PBO

SUMMARY:
The main purpose of this study is to determine if it is safe to use the study drug, clavulanic acid, in combination with cocaine. In this study, subjects will receive intravenous (i.v.) cocaine and the study drug, clavulanic acid. The safety of clavulanic acid is being studied so future studies can be done to find out if this drug is helpful in treating cocaine dependence. Currently, there is no available medication treatment for cocaine dependence.

DETAILED DESCRIPTION:
This is a prospective, placebo controlled inpatient crossover safety study of 3 doses (250 mg/day, 500 mg/day, 750 mg/day) of CLAV with an intravenous infusion of cocaine 40 mg. Subjects will be non-treatment seeking experienced cocaine dependent adults, ages 18-65 (N=12 completers, 21 estimated to enroll). Subjects will undergo a washout of the study drug for 5 half-lives between study drug administration sessions.

The primary objective will be to determine whether there are clinically significant adverse interactions between CLAV (250 mg/day; 500 mg/day; 750 mg/day) and intravenously administered cocaine in healthy, non-treatment seeking adults with cocaine use disorder.

ELIGIBILITY:
Inclusion Criteria:

* Meet Diagnostic and Statistical Manual of Mental Disorders Fifth Edition criteria for cocaine use disorder, moderate to severe.
* Be a non-treatment seeking cocaine user.
* If female and of childbearing potential, must have a negative pregnancy test within 48 hours of beginning the study and be willing to use acceptable contraception or be abstinent for 14 days prior to study, through the entire study and 30 days after study participation.

Exclusion Criteria:

* Be seeking treatment for substance abuse.

(For full inclusion/exclusion criteria or for more information, please contact the site directly.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-10-24 (Actual); Primary Completion 2018-05-25 (Actual); Study Completion 2018-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle M. Kampman, M.D., Principal Investigator — U54 Principal Investigator - University of Pennsylvania; Mary F. Morrison, M.D., M.S., Principal Investigator — Temple University; M. I Walters, M.D., Principal Investigator — Temple University
Locations (1):
- Temple University Hospital - Episcopal Campus, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Uys JD, LaLumiere RT. Glutamate: the new frontier in pharmacotherapy for cocaine addiction. CNS Neurol Disord Drug Targets. 2008 Nov;7(5):482-91. doi: 10.2174/187152708786927868. PMID 19128205
- [Background] Rasmussen BA, Baron DA, Kim JK, Unterwald EM, Rawls SM. beta-Lactam antibiotic produces a sustained reduction in extracellular glutamate in the nucleus accumbens of rats. Amino Acids. 2011 Feb;40(2):761-4. doi: 10.1007/s00726-010-0589-0. Epub 2010 Apr 13. PMID 20383795
- [Background] Ward SJ, Rasmussen BA, Corley G, Henry C, Kim JK, Walker EA, Rawls SM. Beta-lactam antibiotic decreases acquisition of and motivation to respond for cocaine, but not sweet food, in C57Bl/6 mice. Behav Pharmacol. 2011 Aug;22(4):370-3. doi: 10.1097/FBP.0b013e3283473c10. PMID 21543969
- [Background] Kovalevich J, Corley G, Yen W, Rawls SM, Langford D. Cocaine-induced loss of white matter proteins in the adult mouse nucleus accumbens is attenuated by administration of a beta-lactam antibiotic during cocaine withdrawal. Am J Pathol. 2012 Dec;181(6):1921-7. doi: 10.1016/j.ajpath.2012.08.013. Epub 2012 Sep 29. PMID 23031254

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an inpatient study at Temple University, Episcopal Hospital in Philadelphia, Pennsylvania with subjects recruited between 10/24/2016 and 6/04/2018.
Pre-assignment Details: 10 subjects were randomized to one of three treatment arms in a double masked method.
Groups:
- Placebo; Clav 250mg, Then Clav 500mg: Clavulanic acid (Clav) OR Placebo to be given in combination with daily intravenous cocaine; Day #1 IV cocaine only; Day #2: Placebo mg; Day #3: Clav 250 mg; Day #4: Clav 500mg
- Clav 250mg; Placebo; Then Clav 500mg: Clavulanic acid (Clav) OR Placebo to be given in combination with daily intravenous cocaine; Day #2: Clav 250 mg; Day #3: Placebo; Day #4: Clav 500 mg
- Clav 250mg; Clav 500mg; Then Placebo: Clavulanic acid (Clav) OR Placebo to be given in combination with daily intravenous cocaine; Day 1# IV cocaine only; Day #2: Clav 250 mg; Day #3: Clav 500 mg; Day #4: Placebo
Period: IV Cocaine Only (Day 1)
Arm/Group | Placebo; Clav 250mg, Then Clav 500mg | Clav 250mg; Placebo; Then Clav 500mg | Clav 250mg; Clav 500mg; Then Placebo
Started | 3 | 3 | 4
Completed | 3 | 3 | 4
Not Completed | 0 | 0 | 0
Period: FIrst Treatment (Day 2)
Arm/Group | Placebo; Clav 250mg, Then Clav 500mg | Clav 250mg; Placebo; Then Clav 500mg | Clav 250mg; Clav 500mg; Then Placebo
Started | 3 | 3 | 4
Completed | 3 | 3 | 4
Not Completed | 0 | 0 | 0
Period: Second Treatment (Day 3)
Arm/Group | Placebo; Clav 250mg, Then Clav 500mg | Clav 250mg; Placebo; Then Clav 500mg | Clav 250mg; Clav 500mg; Then Placebo
Started | 3 | 3 | 4
Completed | 3 | 3 | 4
Not Completed | 0 | 0 | 0
Period: Third Treatment (Day 4)
Arm/Group | Placebo; Clav 250mg, Then Clav 500mg | Clav 250mg; Placebo; Then Clav 500mg | Clav 250mg; Clav 500mg; Then Placebo
Started | 3 | 3 | 4
Completed | 3 | 3 | 4
Not Completed | 0 | 0 | 0
Period: Added 750mg Dose of CLAV (Day 5)
Arm/Group | Placebo; Clav 250mg, Then Clav 500mg | Clav 250mg; Placebo; Then Clav 500mg | Clav 250mg; Clav 500mg; Then Placebo
Started | 1 (Version 2 of Protocol which added a single blind dose of CLAV 750mg (Period 5) was started after 1 participant had already completed the 4 periods (under Protocol 1) and was discharged. One subject who was enrolled on Protocol version 2 was discontinued before the 750mg dose of CLAV due to an adverse event at a lower dose and never started period 5. Thus, only 1 of the 3 in this arm started period 5.) | 1 (Version 2 of Protocol which added a single blind dose of CLAV 750mg (Period 5) was started after 2 of the subjects in this arm had already completed the 4 periods (under Protocol version 1) and had been discharged. Thus, only 1 subject started Period 5 in this arm.) | 3 (Version 2 of Protocol which added a single blind dose of CLAV 750mg (Period 5) was started after 1 of the participants in this arm had already completed the 4 periods (in protocol 1) and was discharged. Thus, only 3 subjects started Period 5 in this arm.)
Completed | 1 | 1 | 2 (Two of three subjects completed this period. One subject had technical difficulty with IV cocaine infusion resulting in not completed status (Physician decision))
Not Completed | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Clavulanic Acid (CLAV) 250mg, CLAV 500mg Then Placebo (PBO): Clavulanic acid OR Placebo to be given in combination with intravenous cocaine; Day #2: Clavulanic Acid 250 mg (low dose); Day #3: Clavulanic Acid 500 mg; Day #4: Placebo
  Clavulanic acid
  Intravenous cocaine
  Placebo
- CLAV 250mg, PBO, Then CLAV 500mg: Clavulanic acid OR Placebo to be given in combination with intravenous cocaine; Day #2: Clavulanic Acid 250 mg (low dose); Day #3: Placebo; Day #4: Clavulanic Acid 500 mg
  Clavulanic acid
  Intravenous cocaine
  Placebo
- PBO, CLAV 250mg Then CLAV 500mg: Clavulanic acid OR Placebo to be given in combination with intravenous cocaine; Day #2: Placebo; Day #3: Clavulanic Acid 250 mg (low dose); Day #4: Clavulanic Acid 500 mg
  Clavulanic acid
  Intravenous cocaine
  Placebo
- Total: Total of all reporting groups
Arm/Group | Clavulanic Acid (CLAV) 250mg, CLAV 500mg Then Placebo (PBO) | CLAV 250mg, PBO, Then CLAV 500mg | PBO, CLAV 250mg Then CLAV 500mg | Total
Number analyzed (Participants) | 3 | 3 | 4 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 4 | 10
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 50 [46 to 53] | 53 [38 to 60] | 51 [46 to 58] | 51 [38 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 2
  Male | 2 | 3 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 4 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 3 | 8
  White | 0 | 1 | 1 | 2
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 4 | 10
Education Level [Count of Participants; unit: Participants] — Phenotypes and eXposures (PhenX) demographic toolkit. Only number of participants who completed High School/General Educational Development Equivalent or greater are reported
  Participants | 3 | 1 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Severe Adverse Events (AEs)
Description: Rates of occurrence of serious adverse events across the different treatments: Day 1-IV cocaine only; Day 2.3 and 4 treatment with either PBO, CLAV 250mg or CLAV 500mg depending on randomization; Day 5 CLAV 750mg, Day 10 Follow-up appointment
  See Adverse Event section for reporting of mild-moderate AEs.
Time Frame: 6 Days (Study Days 1, 2, 3, 4, 5, 10)
Population: Participants were adults (18-65) with current cocaine use disorder who were recruited from the greater Philadelphia area.
Measure: Count of Participants; unit: Participants
Groups:
- Day 1 - IV Cocaine Only: Subjects received 20mg IV infusion of cocaine and then 40mg IV cocaine at least 2hours 45 minutes after initial infusion
- Placebo (PBO): PBO (followed by IV cocaine given 1 hour (hr) later) was given either on day 2, day 3 or day 4 according to the protocol
- CLAV 250mg: CLAV 250mg (followed by IV cocaine given 1 hr later) was given either on day 2, day 3 or day 4 according to the protocol
- CLAV 500mg: CLAV 500mg (followed by IV cocaine given 1 hr later) was given either on day 2, day 3 or day 4 according to the protocol
- Day 5--CLAV 750mg: CLAV 750mg (followed by IV cocaine given 1 hr later) was given on day 5 according to version 2.3 of the protocol.
- Day 10--Follow up: 5-6 days after discharge, subjects returned for a follow up visit to assess adverse events
Arm/Group | Day 1 - IV Cocaine Only | Placebo (PBO) | CLAV 250mg | CLAV 500mg | Day 5--CLAV 750mg | Day 10--Follow up
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 5 | 10
Participants | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Change in Heart Rate in Response to IV Cocaine Infusion With and Without CLAV Dosing
Description: IV cocaine was infused 1 hour following the dosing of PBO or CLAV 250mg, CLAV 500mg and CLAV 750 mg and vital signs were checked at -15min,-10min, -5 min preinfusion of IV cocaine and then every 2 min for the first 30 minutes, then every 15min through 150 minutes post-infusion. The mean heart rate (HR) at 2 minutes post IV cocaine infusion and the maximum (max) change in heart rate from baseline pre-infusion are reported (peak heart rate post-infusion minus baseline heart rate pre-infusion) are reported.
Time Frame: 4 Days (Study Days 2, 3, 4, 5)
Population: 10 participants were randomized to receive PBO or CLAV 250mg or 500mg on days 2,3 and 4 followed one hour later by IV infusion of cocaine. Part way through the study, a 5th day was added giving CLAV 750mg 1hr before the cocaine infusion (Protocol V2.3). Five participants were eligible for Day 5 but one had technical issues with the cocaine infusion and did not receive the full cocaine dose, so that subject is excluded from the report of day 5 effects.
Measure: Mean (Standard Deviation); unit: beats per minute
Groups:
- Placebo (PBO): Cardiovascular responses to IV cocaine infusion given 1 hour (hr) after PBO (either day 2, day 3 or day 4 according to randomization)
- CLAV 250mg: Cardiovascular responses to IV cocaine infusion given 1 hr after CLAV 250mg (either day 2, day 3 or day 4 according to randomization)
- CLAV 500mg: Cardiovascular responses to IV cocaine infusion given 1 hr after CLAV 500mg (either day 2, day 3 or day 4 according to randomization)
- Day 5--CLAV 750mg: Cardiovascular responses to IV cocaine infusion given 1 hr after CLAV 750mg (day 5 according to version 2.3 of the protocol).
Arm/Group | Placebo (PBO) | CLAV 250mg | CLAV 500mg | Day 5--CLAV 750mg
Number analyzed (Participants) | 10 | 10 | 10 | 4
beats per minute
  HR at 2 min | 82.2 (14.7) | 78.0 (5.7) | 86.8 (13.0) | 91.0 (14.7)
  Max change in HR from baseline | 26.3 (22.6) | 29.8 (19.2) | 32.0 (26.3) | 27.7 (24.7)

3. Primary Outcome: Changes in Blood Pressure in Response to IV Cocaine With and Without CLAV Dosing
Description: IV cocaine was infused 1 hour following the dosing of PBO or CLAV 250mg, CLAV 500mg and CLAV 750 mg and vital signs were checked at -15min,-10min, -5 min pre-infusion of IV cocaine and then every 2 min for the first 30 minutes, then every 15min through 150 minutes post-infusion. The mean systolic blood pressure (SBP) and diastolic blood pressure (DBP) at 2 minutes post IV cocaine infusion are reported. Also, the maximum (max) change in SBP snd DBP from baseline pre-infusion are reported (peak SBP or DBP post-infusion minus baseline SBP or DBP pre-infusion) are reported.
Time Frame: 4 Days (Study Days 2, 3, 4, 5)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo (PBO) | CLAV 250mg | CLAV 500mg | Day 5--CLAV 750mg
Number analyzed (Participants) | 10 | 10 | 10 | 4
mm Hg
  SBP at 2 min | 138.8 (14.8) | 135.0 (15.4) | 140.0 (13.6) | 137.8 (15.5)
  Max change in SBP | 21.6 (13.0) | 23.5 (11.3) | 18.4 (8.9) | 20.9 (16.4)
  DBP at 2 mim | 88.5 (4.6) | 88.8 (11.2) | 89.5 (7.2) | 87.8 (10.0)
  Max change in DBP | 12.1 (2.7) | 13.3 (4.1) | 12.6 (5.1) | 12.7 (3.9)

4. Primary Outcome: Electrocardiogram (ECG) Following IV Cocaine With and Without CLAV Dosing
Description: ECG was done 15 min after IV cocaine infusion (following the dosing of PBO or CLAV 250mg, CLAV 500mg and CLAV 750 mg). The interval between the Q wave and the T wave, corrected (QTc) is reported.
Time Frame: 4 Days (Study Days 2, 3, 4, 5)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Placebo (PBO) | CLAV 250mg | CLAV 500mg | Day 5--CLAV 750mg
Number analyzed (Participants) | 10 | 10 | 10 | 4
ms | 431.8 (16.6) | 432.3 (19.9) | 430.5 (16.3) | 431.3 (14.8)

5. Secondary Outcome: Pharmacokinetic (PK) Parameter of Cocaine-concentration
Description: Cocaine concentrations are reported at 10 min and 30 minutes after cocaine infusion (70 and 90 minutes after administration of placebo (PBO), CLAV 250mg or CLAV 500mg).
Time Frame: 3 Days (Study Days 2, 3, 4)
Population: All 10 participants received PBO, CLAV 250mg or 500mg over 3 days in different order according to randomization. One participant is not included in the analysis due to inadequate samples obtained.
Measure: Mean (Standard Deviation); unit: mg/L
Groups:
- Placebo (PBO) Group-10 Min Cocaine PK: PBO (followed by IV cocaine given 1 hour (hr) later) was given either on day 2, day 3 or day 4 according to the protocol. Cocaine PK level drawn 10 min after IV cocaine infusion (70 min after PBO).
- PBO Group-30 Min Cocaine PK: PBO (followed by IV cocaine given 1 hour (hr) later) was given either on day 2, day 3 or day 4 according to the protocol. Cocaine PK level drawn 30 min after IV cocaine infusion (90 min after PBO).
- CLAV 250mg Group-10 Min Cocaine PK: CLAV 250mg (followed by IV cocaine given 1 hr later) was given either on day 2, day 3 or day 4 according to the protocol. Cocaine PK level drawn 10 min after IV cocaine infusion (70 min after CLAV 250mg).
- CLAV 250mg Group-30 Min Cocaine PK: CLAV 250mg (followed by IV cocaine given 1 hr later) was given either on day 2, day 3 or day 4 according to the protocol. Cocaine PK level drawn 30 min after IV cocaine infusion (90 min after CLAV 250mg).
- CLAV 500mg Group-10 Min Cocaine PK: CLAV 500mg (followed by IV cocaine given 1 hr later) was given either on day 2, day 3 or day 4 according to the protocol. Cocaine PK level drawn 10 min after IV cocaine infusion (70 min after CLAV 500mg).
- CLAV 500mg Group-30 Min Cocaine PK: CLAV 500mg (followed by IV cocaine given 1 hr later) was given either on day 2, day 3 or day 4 according to the protocol. Cocaine PK level drawn 30 min after IV cocaine infusion (90 min after CLAV 500mg)
Arm/Group | Placebo (PBO) Group-10 Min Cocaine PK | PBO Group-30 Min Cocaine PK | CLAV 250mg Group-10 Min Cocaine PK | CLAV 250mg Group-30 Min Cocaine PK | CLAV 500mg Group-10 Min Cocaine PK | CLAV 500mg Group-30 Min Cocaine PK
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9
mg/L | 0.355 (0.111) | 0.240 (0.068) | 0.372 (0.094) | 0.215 (0.046) | 0.344 (0.086) | 0.209 (0.049)

6. Secondary Outcome: Clavulanic Acid (CLAV) Concentrations Following CLAV 250mg and CLAV 500mg Doses
Description: CLAV concentrations were measured 40 min and 70 min after ingestion of CLAV 250 mg or 500 mg. (The 70 min time point is 10 min after the IV cocaine infusion).The 250mg dose and the 500mg dose were given on different days per the randomization protocol: the 250mg dose was given on either day 2 or 3 and the 500mg dose was given on either day 3 or 4.
  The lowest level of detection of CLAV is 40ng/ml. A non-detectable level is reported as 0.
Time Frame: 3 Days (Study Days 2, 3, 4)
Population: 10 subjects received 250mg and 500mg (randomized to different days) but samples for one subject was unusable. A second subject vomited 5 min after both the 250mg dose and the 500mg dose and levels were undetectable; this subject was excluded from analysis. This reports results of 8 subjects.
Measure: Median (Full Range); unit: mg/L
Groups:
- CLAV PK at 250mg Dose--40 Min Time Point: CLAV PK level drawn 40 min after ingestion of CLAV 250 mg
- CLAV PK at 250mg Dose--70 Min Time Point: CLAV PK level drawn 70 min after ingestion of CLAV 250 mg
- CLAV PK at 500mg Dose--40 Min Time Point: CLAV PK level drawn 40 min after ingestion of CLAV 500 mg
- CLAV PK at 500mg Dose--70 Min Time Point: CLAV PK level drawn 70 min after ingestion of CLAV 500 mg
Arm/Group | CLAV PK at 250mg Dose--40 Min Time Point | CLAV PK at 250mg Dose--70 Min Time Point | CLAV PK at 500mg Dose--40 Min Time Point | CLAV PK at 500mg Dose--70 Min Time Point
Number analyzed (Participants) | 8 | 8 | 8 | 8
mg/L | 0.036 [0 to 4.015] | 0.506 [0 to 4.000] | 0.394 [0 to 1.993] | 1.912 [0.181 to 3.940]

7. Secondary Outcome: Difference in CLAV Concentrations Between the 250mg and 500mg CLAV Doses
Description: The CLAV concentration after ingestion of 250mg CLAV minus the CLAV PK level after the 500 mg dose is reported at 40min and 70 min after ingestion
Time Frame: 3 days (Day 2, 3, 4)
Population: 10 subjects were randomized and received 250mg and 500mg on different days based on their randomization. One subject's samples were unusable. A second subject vomited after each dose (250mg and 500mg), had nondetectable levels and was excluded in the calculation. This analysis is based on 8 subjects.
Measure: Median (Full Range); unit: mg/L
Groups:
- 40 Minute Time Point After 250mg CLAV vs. 500mg CLAV: CLAV PK level 40 minutes after ingestion of CLAV 250mg minus the CLAV PK level 40 minutes after ingestion of CLAV 500mg
- 70 Minute Time Point After 250mg CLAV vs. 500mg CLAV: CLAV PK level 70 minutes after ingestion of CLAV 250mg minus the CLAV PK level 70 minutes after ingestion of CLAV 500mg
Arm/Group | 40 Minute Time Point After 250mg CLAV vs. 500mg CLAV | 70 Minute Time Point After 250mg CLAV vs. 500mg CLAV
Number analyzed (Participants) | 8 | 8
mg/L | 0.227 [-2.022 to 1.405] | 0.331 [-2.944 to 2.800]
Statistical Analysis 1: Comparison: 40 Minute Time Point After 250mg CLAV vs. 500mg CLAV; Test type: Superiority; p = 0.69, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: 70 Minute Time Point After 250mg CLAV vs. 500mg CLAV; Test type: Superiority; p = 0.46, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Pupil Pharmacodynamic Effects of Cocaine With Clavulanic Acid
Description: Pupil Diameter (mm) was measured 10 minutes pre-infusion and 10, 15, 30 and 45 min after cocaine infusion. Cocaine infusion was done 1 hour following ingestion of placebo (day 2), CLAV 250 mg (day3), or CLAV 500 mg (day 4). Results are reported as median pupil diameter (mm) with interquartile range at different time points relative to the cocaine infusion as noted.
Time Frame: 10 minutes pre-infusion and 10, 15, 30 and 45 min after cocaine infusion on Study Days 2, 3, and 4
Population: 10 subjects receiving IV cocaine infusion were randomized to receive either PBO, CLAV 250mg or CLAV 500mg on days 2, 3,and 4 depending on randomization
Measure: Median (Inter-Quartile Range); unit: mm
Groups:
- Placebo (PBO): Pupil diameter response to IV cocaine infusion given 1 hour (hr) after PBO (either day 2, day 3 or day 4 according to randomization)
- CLAV 250mg: Pupil diameter responses to IV cocaine infusion given 1 hr after CLAV 250mg (either day 2, day 3 or day 4 according to randomization)
Arm/Group | Placebo (PBO) | CLAV 250mg | CLAV 500mg
Number analyzed (Participants) | 10 | 10 | 10
mm
  -10 min pre-infusion | 3.1 [2.8 to 3.5] | 3.10 [2.7 to 3.4] | 3.20 [2.8 to 3.5]
  10 min post-infusion | 3.55 [3.3 to 3.9] | 3.70 [3.5 to 4.5] | 3.90 [3.6 to 4.5]
  15 min post-infusion | 3.55 [3.3 to 3.7] | 3.40 [3.0 to 4.3] | 3.50 [3.2 to 4.1]
  30 min post-infusion | 3.6 [3.2 to 4.1] | 3.30 [2.9 to 4.1] | 3.35 [3.0 to 4.1]
  45 min post-infusion | 3.4 [3.2 to 4.0] | 3.10 [2.8 to 3.6] | 3.10 [2.7 to 3.7]

ADVERSE EVENTS:
Time Frame: Adverse Event Data was systematically collected daily during the 5 or 6 day inpatient period and up to their follow up visit at day 10. Any subjects who continued to experience adverse events after the follow up visit were followed until all adverse events resolved.
Description: Participants were evaluated daily by a physician for adverse events, and had 24 hour access to medical staff during the inpatient period to report adverse events.
Groups:
- Day 1-IV Cocaine Infusion Only: Subjects received IV cocaine 20mg and then at least 2hr 45min later they received IV cocaine 40mg
- Placebo + IV Cocaine: Subjects were randomized to receive oral matched placebo (on day 2, 3 or 4) followed by IV cocaine 40mg 1hr later
- CLAV 250mg + IV Cocaine: Subjects were randomized to receive oral CLAV 250mg (on day 2, 3 or 4) followed by IV cocaine 40mg 1hr later
- CLAV 500mg + IV Cocaine: Subjects were randomized to receive oral CLAV 500mg (on day 2, 3 or 4) followed by IV cocaine 40mg 1hr later
- Day 5--CLAV 750mg + IV Cocaine: Protocol V2.3 allowed for subjects to proceed to day 5 receiving 750mg after they completed Day 2,3 and 4 and received PBO, CLAV 250mg and CLAV 500mg iper day n some randomized order
- Discharge Day: Day after last dose of study drug (Day 6 for those completing day 5 CLAV 750mg; ot Day 5 for those completing days 1-4 only)
- Day 10-Follow-up: All subjects returned for a follow-up visit on Day 10 of the study (5-6 days after discharge)
Arm/Group | Day 1-IV Cocaine Infusion Only | Placebo + IV Cocaine | CLAV 250mg + IV Cocaine | CLAV 500mg + IV Cocaine | Day 5--CLAV 750mg + IV Cocaine | Discharge Day | Day 10-Follow-up
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/5 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/5 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 5/10 | 4/10 | 3/10 | 3/10 | 2/5 | 5/10 | 4/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Day 1-IV Cocaine Infusion Only (N=10) | Placebo + IV Cocaine (N=10) | CLAV 250mg + IV Cocaine (N=10) | CLAV 500mg + IV Cocaine (N=10) | Day 5--CLAV 750mg + IV Cocaine (N=5) | Discharge Day (N=10) | Day 10-Follow-up (N=10)
upper respiratory infection (URI) (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2) — one with upper respiratory infection; one with flu
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 — Two occurrences in one subject: 3 consecutive ventricular complexes on day 1 and 4 consecutive beats ventricular complexes on day of CLAV 500mg dose
Abdominal gas (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 | 0 | 1 (1) | 0 — 3 events in 2 subjects; one subject had event on day 1 and CLAV 250mg day. The 2nd subject's event was on discharge day
Nausea+vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 | 0 | 0 — 2 events in 1 subject--after CLAV 250mg and CLAV 500mg
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Indigestion (Gastrointestinal disorders) | 0 | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0
Reaction to Telemetry Pads on Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Itchy Skin (Skin and subcutaneous tissue disorders) | 0 | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 — Itchiness was located near IV injection site
Teary eyes (Eye disorders) | 1 (2) | 0 | 1 (1) | 0 | 0 | 0 | 0
Lower eyelid twitch rhythmic (Eye disorders) | 1 (1) | 0 | 0 (0) | 0 | 0 | 0 | 0 — Right eye only
Elevated calcium levels (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 | 0 | 0
Hand bilateral spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 1 (1)
Lightheaded (Nervous system disorders) | 1 (2) | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 — 1 subject, 4 events
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 — 3 subject, 4 events; one subject had headache on day 5 (CLAV 750mg) and day 6 (discharge day)
Drowsiness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0
Insomnia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0
Tooth Ache (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 1 (1) | 0
hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0

LIMITATIONS AND CAVEATS:
The sample size was relatively small (n=10) and the current study was not powered to adequately explore efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results in this trial are considered proprietary and still under evaluation.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-22): https://cdn.clinicaltrials.gov/large-docs/69/NCT02563769/Prot_SAP_000.pdf